CLINICAL TRIAL: NCT05912088
Title: Effectiveness of the sLiFE Program to Reduce Falls and Frailty in Elderly People in Primary Care. Randomized Clinical Trial
Brief Title: Elderly Falls Prevention With sLiFE Program in Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GRS 2502/B/22
Record Dates: First submitted 2023-06-11; First posted 2023-06-22 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-06

CONDITIONS: Accidental Falls; Frailty; Elderly; Activities, Motor
MeSH Terms: conditions — Frailty; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The strength and balance activities of the sLiFE program will be carried out. Participants will be invited to participate in groups of about 14 people in Primary Care Heath Centers.
  Interventions: Behavioral: Intervention Group
- Control Group (Placebo Comparator): Participants will receive the usual health advice.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Intervention Group — Subjects will participate in groups of about 14 to implement the program.
  Arms: Intervention Group
Behavioral: Control Group — Subjects will receive the usual care advice
  Arms: Control Group

SUMMARY:
This study aims to guide older people living in the community on appropriate strategies within a fall prevention program. This program is aimed at training in daily activities carried out through group workshops (guided by a physiotherapist) and at preventing risk situations at home.

DETAILED DESCRIPTION:
Two-arm, non-blind, non-inferiority experimental design. Multicenter, randomized trial.

The study tries to assess whether a group intervention following the principles of the sLiFE program is more effective than an usual health advice reducing the incidence of falls.

ELIGIBILITY:
Inclusion Criteria:

* People older than 65 years of age
* Living at home
* Speak and read Spanish

Exclusion Criteria:

* Heart failure (NYHA class III and IV)
* Recent stroke (<6 months)
* Parkinson's disease
* In active cancer treatment (last 6 months)
* GOLD class III and IV chronic obstructive pulmonary disease
* Unstable lower extremity fracture
* Amputated lower extremity
* Treatment less than 6 months of depression
* Uncontrolled resting blood pressure of a systolic > 160 or diastolic > 100 or more
* Unavailability for intervention, planned travel or relocation more than 2 months within the first 6 months of the study
* Moderate to severe cognitive impairment (Mini Mental cognitive assessment <23)
* Current participation in another interventional clinical trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of falls | 6 months
  Number of falls in relation to the degree of physical activity.
Physical activity | 8 days
  It will be evaluated with a digital pedometer for 9 consecutive days
Physical activity | 6 months
  It will be evaluated with the Global Physical Activity Questionnaire
Frailty | 6 months
  Frailty will be measured according to the five criteria of Fried's phenotype: 1) Low muscle strength; 2) Poor nutrition; 3) Poor endurance; 4) Slow walking and 5) Low physical activity.
Health effects | 6 months
  It will be measured using the quality of life questionnaire EQ-5D

SECONDARY OUTCOMES:
Fear of falling | 6 months
  It will be assesses using the Short Falls International Scale of Efficacy (Short FES I). It measures of "concerns about falling". This scale has 7 items with a Likert scale with 4 options: 1) not at all concerned, 2) somewhat concerned, 3) fairly concerned, and 4) very concerned.
Cognitive assessment | 6 months
  It will be evaluated with the Montreal Cognitive Assessment (MoCA): 30 questions and takes 10-12 minutes to complete.
Motor function | 6 months
  It will be evaluated with the Short Physical Performance Battery (SPPB). It assesses three aspects of mobility: balance, gait speed and strength of limbs or lower limbs to get up from a chair
Adherence to exercise | 6 months
  It will be assessed using the Exercise Adherence Rating Scale (EARS). It is composed of 16 items scored using a 5-point Likert scale (0 = completely agree to 4 = completely disagree) with a possible summed score range from 0 to 64.

CONTACTS AND LOCATIONS:
Overall Officials: Luis García-Ortiz, Dr, Study Chair — Primary Health Care Research Unit
Locations (1):
- Primary Care Research Unit of Salamanca (APISAL), Salamanca, Spain

REFERENCES:
- [Derived] Llamas-Ramos I, Llamas-Ramos R, Lugones-Sanchez C, Gonzalez-Garcia S, Tamayo-Morales O, Alvarado-Omenat JJ, Pablos-Hernandez C, Gomez-Marcos MA, Garcia-Ortiz L, Rodriguez-Sanchez E. Effect of a lifestyle-integrated functional exercise (LiFE) group intervention (sLiFE) to falls prevention in non-institutionalized older adults. Protocol of a randomised clinical trial. Front Public Health. 2024 Jan 8;11:1304982. doi: 10.3389/fpubh.2023.1304982. eCollection 2023. PMID 38259747